CLINICAL TRIAL: NCT03507361
Title: Heart Rate Variability-based Music for the Prevention of PCI-related Myocardial Injury
Brief Title: Myocardial Damage and Music Study
Acronym: MYDA-MUSIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Filippo Neri General Hospital (Other)
Responsible Party: Principal Investigator, Christian Pristipino, Principal investigator, San Filippo Neri General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V1-Jan31-2018
Record Dates: First submitted 2018-03-26; First posted 2018-04-25 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Chronic Stable Angina; PTCA
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC (Experimental): Music will be administered through a normal computer equipped with a technology (Sound-of-Soul) that translates the patient's heart rate variability (HRV) into sounds according to a digital computer music-library. Music will start 10 minutes before and will end at the completion of the interventional procedure
  Interventions: Other: HRV-BASED MUSIC
- DUMB EARPHONES (No Intervention): Dumb earphones will be placed over patient's ears starting 10 minutes before and ending at the completion of the interventional procedure.

INTERVENTIONS:
Other: HRV-BASED MUSIC — Music is produced by Sound-of-Soul technology that translates HRV power frequency spectrum real-time into music. The intervals between the heartbeats are detected in milliseconds and then transferred into a frequency spectrum. Sound of Soul system gets wired into different band pass filters which are linked to the frequencies of the heart (i.e. low frequency and high frequency). Once the signal is detected and computed, the Sound of Soul system links it through a musical instrument digital interface (MIDI). This interface transforms ECG data into music and sounds. The audio production is performed using a virtual instrumentation technology with different music libraries. For the puropose of this study, all patients will ear the same instrument (arp). Once the instrument have been selected, the ECG gets recorded and in real-time the patient can hear a music obtained from his/her own HRV. The investigator will control the volume and the different settings of the music.
  Arms: MUSIC

SUMMARY:
MYDA-MUSIC study is a randomized, double blind (operator and analyst) study performed in San Filippo Neri Hospital, Roma, Italy and in Di Venere Hospital, Bari, Italy. The planned study duration is 12 months. The objectives are to assess the effects of heart-rate-variability based music on the incidence and magnitude of peri-procedural myocardial damage caused by coronary angioplasty in stable patients. 443 patients with chronic stable angina scheduled for a coronary angiography and possible ad hoc angioplasty will be randomized to receive music or dumb earphones.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stable angina scheduled to undergo a coronary angiography and ad-hoc angioplasty

Exclusion Criteria:

* Abnormal c-TnI level before angiography
* Participation in other clinical studies
* Patients with pacemakers or defibrillators
* High rate atrial fibrillation (baseline heart rate >99 bpm) at enrolment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure-related myocardial injury | within 24 hours from interventional procedure
  c-TnI concentration >99th percentile URL in at least 1/3 blood drawings

SECONDARY OUTCOMES:
Overall satisfaction with the procedure | From 5 to 30 minutes after the interventional procedure
  Self-evaluation test on an analogic visual scale (score range 1-10, higher stress for higher values)
Difference in Distress self-evaluation baseline and after the intervention | Baseline and from 5 to 30 minutes after the interventional procedure
  Self-evaluation test on an analogic visual scale (score range 1-10, higher stress for higher values)
Evaluation of pain experienced during the interventional procedure | Baseline and from 5 to 30 minutes after the interventional procedure
  Self-evaluation test (score range 1-10, higher pain for higher values)
Difference in Anxiety evaluation baseline and after the intervention | Baseline and from 5 to 30 minutes after the interventional procedure
  State-Trait Anxiety Inventory (STAI) test - Y italian version (score range 20-80, the higher the score the more anxiety the patients has, 2 subscales)
Questionnaire regarding a narrative report of the procedure | From 5 to 30 minutes after the interventional procedure
  Categorical analysis evaluated with a dedicated software analysing unstructured written narration of the experience of their invasive procedure.
Changes in Mean Heart rate during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (recorded for 5 to 10 minutes)
  Calculation of Mean HR (beats/minute) on ECG samples recorded for 5 to 10 minutes
Changes in RR during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of Mean RR interval (msec) on 5 to 10 minutes duration ECG samples.
Changes in SDNN during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of SDNN (msec) on 5 to 10 minutes duration ECG samples.
Changes in RMSSD during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of RMSSD (msec) on 5 to 10 minutes duration ECG samples.
Changes in pNN50 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of pNN50 (%) on 5 to 10 minutes duration ECG samples.
Changes in pNN20 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of pNN20 (%) on 5 to 10 minutes duration ECG samples.
Changes in pNN10 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of pNN10 (%) on 5 to 10 minutes duration ECG samples.
Changes in pNN05 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of pNN05 (%) on 5 to 10 minutes duration ECG samples.
Changes in SD1 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of SD1 (msec) on 5 to 10 minutes duration ECG samples.
Changes in SD2 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of SD2 (msec) on 5 to 10 minutes duration ECG samples.
Changes in SD1/SD2 during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of SD1/SD2 ratio (number) on 5 to 10 minutes duration ECG samples.
Changes in VB during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of VB (sec) on 5 to 10 minutes duration ECG samples.
Changes in Stress index during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of stress index (number) on 5 to 10 minutes duration ECG samples.
Changes in CV during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of CV (number) on 5 to 10 minutes duration ECG samples.
Changes in Power of frequency domains during the procedure (Heart rate variability measure) | Baseline and at 5 minutes intervals (5 to 10 minutes duration)
  Calculation of the power of VLF, LF, HF and total frequency-domain power on 5 to 10 minutes duration ECG samples (ms2)
Postprocedural c-TnI peak concentration in patients undergoing coronary angioplasty | within 24 hours from interventional procedure
  Highest concentration in c-TnI in 3 blood samples
Time-to-peak in c-TnI concentration in patients undergoing coronary angioplasty | within 24 hours from interventional procedure
  Time-to-Highest concentration in c-TnI in 3 blood samples
Incidence of procedure-related myocardial infarction (myocardial infarction type 4a) in patients undergoing coronary angioplasty | within 24 hours from interventional procedure
  c-TnI concentration >10 x the 99th percentile in at least 1/3 blood drawings
Incidence of in-hospital Major Adverse Cardiac Events in patients undergoing coronary angioplasty | Through study completion (average of 3 days)
  Incidence of death, myocardial infarction, unplanned revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- San Filippo Neri General Hospital, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided